CLINICAL TRIAL: NCT00629603
Title: Polymorphisms of Fibrosis-Relating Genes on Outcome of HCV-Related Chronic Liver Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Principal Investigator, Jung-Fa,Tsai (1), Professor of Medicine, Kaohsiung Medical University Chung-Ho Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: KMUH-IRB-950347
Record Dates: First submitted 2008-02-26; First posted 2008-03-06 (Estimated); Last update posted 2013-04-18 (Estimated); Status verified 2013-04

CONDITIONS: Fibrosis; Chronic Liver Disease
Keywords: hepatitis C virus infection; chronic liver disease; fibrosis-related cytokine
MeSH Terms: conditions — Fibrosis; Hepatitis C | interventions — Cytokines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cytokine polymorphisms, HCV infection (Experimental): Relate the fibrosis cytokine gene polymorphisms with disease severity of HCV-related chronic liver disease
  Interventions: Genetic: cytokine; Genetic: cytokine polymorphisms; Genetic: cytokine polymorphism

INTERVENTIONS:
Genetic: cytokine — polymorphisms of fibrosis-relating cytokine were measured to validate the effectiveness of fibrosis in HCV-related chronic liver disease
  Other Names: hepatitis C virus infection; cytokine polymorphism; fibrosis
Genetic: cytokine polymorphisms — Fibrosis-relating cytokine polymorphisms in hepatitis C virus-related chronic liver disease were measured to validate the degree of fibrosis
  Other Names: hepatitis C virus infection; cytokine polymorphism; fibrosis
Genetic: cytokine polymorphism — fibrosis-relating cytokine polymorphism
  Other Names: hepatitis C virus infection; cytoline polymorphism; fibrosis

SUMMARY:
Hepatitis C virus (HCV) infection causes different disease spectrum ranging from minimal progressive liver disease to cirrhosis or hepatocellular carcinoma. Evidence indicates that host genetic factor may play a role in determining disease progression. It is known that many cytokine polymorphisms affect disease progressin via increasing hepatic fibrosis that are key factors in progressing liver injury. By combinations of fibrosis-relating gene polymorphisms, this study aims to identify patients with high risk for progressive liver disease. These patients need intensive therapy to decrease morbidity and mortality of chronic HCV-related liver disease.

DETAILED DESCRIPTION:
Determination of the following fibrosis-relating gene polymorphisms in HCV-related chronic liver disease and HCC will be performed: TNF-α , TNF-β, Factor V Leiden, TGF-β1, PDGF-B gene, Angiotensinogen (AT),Angiotensin converting enzyme (ACE), microsomal epoxide hydrolase (mEH) and glutathione-S-transferase (GST).

ELIGIBILITY:
Inclusion Criteria:

* Patients with anti-HCV positive

Exclusion Criteria:

* Anti-HCV-negative patients

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2007-01; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
cytokine gene polymorphism on disease severity | years

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Fa Tsai, M.D., Ph.D., Principal Investigator — Professor of Medicine
Locations (2):
- Taiwan (2):
  - Kaohsiung Medical University Chung-Ho Hospital, Kaohsiung City, Kaohsiung
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Kaohsiung